CLINICAL TRIAL: NCT01733277
Title: A Cross-sectional Study to Explore the Osteoarthritis Structural Changes Assessed by MRI That Are Biomarkers of Neuropathic Pain in Knee Osteoarthritis
Brief Title: Osteoarthritis Structural Changes Assessed by Magnetic Resonance Imaging and Neuropathic Pain in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: ArthroLab Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A122-MER12H
Record Dates: First submitted 2012-11-16; First posted 2012-11-27 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-05

CONDITIONS: Neuropathic Pain; Knee Osteoarthritis
Keywords: Neuropathic pain; Knee osteoarthritis; MRI
MeSH Terms: conditions — Neuralgia; Osteoarthritis, Knee | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With neuropathic pain (PainDETECT ≥ 13): Magnetic Resonance Imaging (MRI)
  Interventions: Other: Magnetic Resonance Imaging (MRI)
- No neuropathic pain (PainDETECT<13): Magnetic Resonance Imaging (MRI)
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — All participants from both arms will be subjected to MRI

SUMMARY:
The primary objective of this study is to identify osteoarthritis (OA) structural changes, as assessed by MRI, that best correlate with the presence of neuropathic pain (NP) using the PainDETECT questionnaire (PainDETECT ≥ 13) on a population of patients with OA of the knee experiencing moderate to severe pain (VAS ≥ 40 mm).

DETAILED DESCRIPTION:
This study is a multicentre, cross-sectional observational pilot study. The presence of NP was determined based on use of the PainDETECT questionnaire (score 1 to 38), the score of which was defined for the purpose of the study as ≥ 13. A total of 50 OA patients with moderate to severe pain (VAS ≥ 40), 25 without the presence of NP (OA/NP-) (PainDETECT score < 13), and 25 with the presence of NP (OA/NP+) (PainDETECT score ≥ 13) were enrolled. Since this is a pilot study, we arbitrarily determined the number of patients at 50, which represents 25 patients per arm, a number deemed sufficient to identify the knee OA structural changes that could be preferentially associated with NP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either sex, aged 40 years and more;
* Followed in an ambulatory clinic;
* Presenting with primary OA of the knee according to American College of Rheumatology (ACR) criteria;
* With an OA of radiological stages 2 and 3 according to Kellgren-Lawrence;
* Knee pain for at least 1 month out of the 3 months preceding the study;
* Visual Analog Scale (VAS) of pain while walking on a flat surface ≥ 40 mm;
* Agrees to sign the Informed Consent Form;
* Not taking part in another clinical trial;
* Agrees to respect the protocol.

Exclusion Criteria:

* Other bone and articular diseases (antecedents and/or current signs);
* Presenting with isolated knee lateral compartment OA defined by joint space loss in the lateral compartment only;
* Knee surgery on the study knee;
* Comorbidities that restrict knee function;
* Had received any investigational drug within 30 days or 5 half lives (whichever is greater) prior to entering the study;
* Unable to give informed consent;
* Counter-indication to an MRI examination;
* Baseline Visit cartilage volume cannot be calculated from the MRI due to advanced OA or any other technical reason;
* Abnormal findings and or any other condition, which, in the Investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data through MRI to achieve the objectives of the study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presence or absence of neuropathic pain on a population of patients with OA of the knee experiencing moderate to severe pain (VAS ≥ 40 mm)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Raynauld, MD, Principal Investigator — Université de Montréal
Locations (2):
- Canada (2):
  - Institut de Rhumatologie de Montréal, Montreal, Quebec
  - Centre de Rhumatologie St. Louis, Québec, Quebec

REFERENCES:
- [Derived] Roubille C, Raynauld JP, Abram F, Paiement P, Dorais M, Delorme P, Bessette L, Beaulieu AD, Martel-Pelletier J, Pelletier JP. The presence of meniscal lesions is a strong predictor of neuropathic pain in symptomatic knee osteoarthritis: a cross-sectional pilot study. Arthritis Res Ther. 2014 Dec 14;16(6):507. doi: 10.1186/s13075-014-0507-z. PMID 25497320

RESULTS

PARTICIPANT FLOW:
Groups:
- Presence of Neuropathic Pain: Presence of neuropathic pain using the PainDETECT questionnaire (PainDETECT ≥ 13)
  MRI
- Absence of Neuropathic Pain: Absence of neuropathic pain using the PainDETECT questionnaire (PainDETECT < 13)
  MRI
Period: Overall Study
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Number; unit: participants]
  40-90 years | 25 | 25 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 50
PainDetect (0-38) [Mean (Standard Deviation); unit: units on a scale] — The presence of neuropathic was determined based on use of PainDETECT questionnaire which can discriminate patients with neuropathic knee pain (score ≥ 13; the higher the score, the worst is the pain).
  units on a scale | 21.1 (5.4) | 8.1 (2.6) | 14.6 (7.8)
VAS Pain (0-100) [Mean (Standard Deviation); unit: units on a scale] — Visual Analogue Scale (VAS) for global knee pain (0 mm = no pain, 100 mm = most severe pain)
  units on a scale | 67 (13) | 62 (14) | 64 (13)

OUTCOME MEASURES:

1. Primary Outcome: Osteoarthritis Structural Changes Assessed by Quantitative Magnetic Resonance Imaging With and Without Neuropathic Pain
Time Frame: Baseline
Population: Number of participant analyzed Per-protocol
Measure: Number; unit: participants
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain
Number analyzed (Participants) | 25 | 25
participants
  Partial Meniscal Extrusion (Medial) | 14 | 7
  Partial Meniscal Extrusion (Lateral) | 5 | 1
  Bone Marrow Lesions (Lateral Plateau) | 15 | 8

2. Secondary Outcome: Variation in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores (Total, Pain, Function, Stiffness) and the Presence or Absence of Neuropathic Pain
Description: The WOMAC measures pain (score range 0-20), stiffness (score range 0-8), and functional limitation (score range 0-68) for a Total (cumulative score range 0-96) where the higher the score the worst the pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain
Number analyzed (Participants) | 25 | 25
units on a scale
  WOMAC (total: 0-96) | 62 (15) | 45 (21)
  WOMAC (Pain: 0-20) | 59 (15) | 43 (17)
  WOMAC (Stiffness: 0-8) | 62 (19) | 51 (24)
  WOMAC (Function: 0-68) | 62 (16) | 45 (23)

3. Other Pre Specified Outcome: Correlation Between the Presence of Neuropathic Pain and Biological Marker of Inflammation (CRP)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain
Number analyzed (Participants) | 25 | 25
mg/L | 5.7 (6.6) | 4.3 (2.9)

ADVERSE EVENTS:
Arm/Group | Presence of Neuropathic Pain | Absence of Neuropathic Pain
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No